CLINICAL TRIAL: NCT02512653
Title: Biological Standarization of Cupressus Arizonica Allergen Extract to Determine the Biological Activity in Histamine Equivalent Units (HEP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 608-PR-PRI-199
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Allergy to Tree Pollen
Keywords: Allergy to Cupressus pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cupressus arizonica allergen extract at 4 different concentrations. Positive control. Negative control
  Interventions: Biological: Cupressus arizonica

INTERVENTIONS:
Biological: Cupressus arizonica — Four different concentrations of Cupressus arizonica allergen extract, positive control and negative control

SUMMARY:
Biological Standardization of Cupressus arizonica Allergen Extract.

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent, appropriately signed and dated by subject.
* Subject can be male or female of any race and ethinic group.
* Age 18 years and 60 years ata the study inclusión day.
* Positive clinical history of inhalatory allergy to Cupressus arizonica.
* A positive prick test with a standarices commercially Cupressus arizonica allergen extract.
* A positive prick test with positive control of histamine 10 mg/ml.
* A positive test for specific IgE to Cupressus arizonica.

Exclusion Criteria:

* Immunotherapy in the past 5 years with an allergen extract Cupressus arizonca or other allergen extract than may interfere with the allergene to be tested.
* Use of drugs that may interfere before and after with the skin reactions.
* Treatment with certain drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the inmediate phase | Test sites should be inspected and recorded 15-20 min after application

CONTACTS AND LOCATIONS:
Overall Officials: Lena Erbiti, Study Chair — Laboratorios Leti, S.L.U
Locations (2):
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Fuenalabrada, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid